CLINICAL TRIAL: NCT00331331
Title: The Vitreous Proteome and Inflammatory Mediators in Ocular Inflammatory Disease
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060068; 06-EI-0068
Record Dates: First submitted 2006-05-27; First posted 2006-05-29 (Estimated); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Uveitis; Vasculitis; Ocular Inflammatory Disease
Keywords: Uveitis; Intermediate Uveitis; OCULAR INFLAMMATORY DISEASE; Macular Edema; Vasculitis; Natural History
MeSH Terms: conditions — Uveitis; Vasculitis; Uveitis, Intermediate; Macular Edema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Vitreous, anterior chamber fluid, whole blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Participants with appropriate ocular disorders who were previously enrolled as part of the MUST study and patients who participate in other intramural NIH studies

SUMMARY:
This study will examine the proteins of people with uveitis, or inflammation of the eyes. Evaluating the vitreous, the colorless transparent substance that fills the eyeball in back of the lens, is now possible with the use of new microtechnology. There is an opportunity to evaluate the kinds of proteins that are present in severe, noninfectious sight-threatening uveitis.

Up to 300 participants, ages 18 and older with the appropriate ocular disorders and where vitreous or anterior chamber fluid specimens can be obtained, will be enrolled in the study. This number includes participants that were previously enrolled as part of the Multicenter Uveitis Steroid Treatment (MUST) study, as well as patients who participate in other intramural NIH studies and agree to participate in this study. Researchers will study the vitreous that will be removed from patients' eyes during an operation to insert a steroid implant. The steroid implant is used instead of immunosuppressive therapy, a way to reduce the action of the immune system.

Patients will undergo a procedure involving a small hole made in the eye into which the implant is placed. Normally a small amount of the vitreous comes out during that procedure, and in this study, the vitreous specimen will be taken for testing of inflammatory products. At the same time, a small sample of blood, about 1-1/2 tablespoons, will be collected so that the researchers can compare inflammatory products that may be in the blood with those in the vitreous. If a patient needs to have the implant placed again during the study, he or she would be asked permission for collection of the vitreous and blood samples, as previously. Samples collected will not be used to diagnose patients' conditions or to change any treatments being done. All samples will be labeled with special code numbers so that there is no identifying information about patients. This study will not involve examinations or scheduled visits of patients.

DETAILED DESCRIPTION:
Newer therapies to treat many ocular disorders including uveitis are being considered and studied. We do not have a clear picture as to what lymphokines/chemokines are present in the vitreous or anterior chamber fluid of patients with active intraocular inflammatory disease as well as other disorders with a proposed inflammatory component such as age-related macular degeneration (AMD) and diabetes. Further, no studies have been yet performed evaluating the proteome of the vitreous or anterior chamber fluid in the uveitic, AMD and diabetic state.

This is a natural history study with specimens taken after indicated surgery for patients with uveitis and other studies. Specimens of anterior chamber fluid and vitreous will be evaluated for 32 cytokines and the proteome using systems permitting the evaluation of small amounts of material. A serum sample will be taken at the same time to compare with the lymphokine profile found in the vitreous. Previously, patients participating in the MUST (Multicenter Uveitis Steroid Treatment) study, a randomized study evaluating an ocular steroid implant versus standard immunosuppressive therapy for the treatment of intermediate and posterior uveitis, were enrolled. However, as the MUST study is complete; we are currently only accepting participants from the NEI or other intramural NIH studies where permission is obtained from the patient to allow such evaluations to be done.

ELIGIBILITY:
INCLUSION CRITERIA:

Participants must participate in a study that permits the evaluation of specimens.

EXCLUSION CRITERIA:

Eligible participants who do not wish to donate their vitreous specimen or anterior chamber fluid, as appropriate, or blood sample or undergo a blood draw for the purposes of this research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 300 participants will be enrolled in the study. This number includes participants that were previously enrolled as part of the MUST study, as well as patients who participate in other intramural NIH studies and agree to participate in this study. The MUST study collection has been completed and this study is open to all qualifying participants.
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2007-02-14 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
To compare the vitreous and anterior chamber fluid immune/protein profile with that of the peripheral blood. | duration of the study
  To compare the vitreous and anterior chamber fluid immune/protein profile with that of the peripheral blood.
To begin to develop a proteomic picture of the vitreous and anterior chamber fluid. | duration of study
  To begin to develop a proteomic picture of the vitreous and anterior chamber fluid.
To gather information about the kinds of cytokines/lymphokines, biomarkers, proteome and exosomes that are present in the vitreous and AC fluid of an eye with uveitis as well as other retinal disorders such as AMD, diabetes and others. | duration of the study
  To gather information about the kinds of cytokines/lymphokines, biomarkers, proteome and exosomes that are present in the vitreous and AC fluid of an eye with uveitis as well as other retinal disorders such as AMD, diabetes and others.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Y Chew, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2006-EI-0068.html